CLINICAL TRIAL: NCT00874640
Title: Patient Characteristics in Daily Radiological Practice of Gadovist® Application (PATRON)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14317; GV0810DE (Other: Company internal)
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Epidemiologic Factors
Keywords: Drug utilization review
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Biological: Gadobutrol (Gadovist, BAY86-4875) — Patients with indication for a MRT or MR-Angiography and for whom the radiologist has decided to use the contrast medium gadobutrol

SUMMARY:
To evaluate patient characteristics in the current daily radiological practice of Gadovist application. Special focus will be laid on the individual risk factors of patients, the indications for and the dose of Gadovist application.

Secondary objective is to prove the known safety profile (especially rare adverse events) of Gadovist and to collect data on handling problems with different application forms (one questionnaire per center).

ELIGIBILITY:
Inclusion Criteria:

* patients with indication for a MRT or MR-Angiography and for whom the radiologist has decided to use the contrast medium Gadovist

Exclusion Criteria:

* No exclusion criteria besides the contraindications for the use of Gadovist as mentioned in the German product information.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Radiological practice
Sampling Method: Non-Probability Sample
Enrollment: 3711 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Patient Profile | At day of application

SECONDARY OUTCOMES:
Dosing of Gadovist in different indications | At time of application
Adverse Events | Throughout and after application

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany